CLINICAL TRIAL: NCT02504892
Title: Phase 2 Study of Everolimus Therapy in Patients With Birt-Hogg-Dube Syndrome (BHD)-Associated Kidney Cancer or Sporadic Chromophobe Renal Cancer
Brief Title: Everolimus Therapy in People With Birt-Hogg-Dube Syndrome (BHD)-Associated Kidney Cancer or Sporadic Chromophobe Renal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to slow, insufficient accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ramaprasad Srinivasan, M.D., Principla Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 150166; 15-C-0166
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Results first posted 2019-03-07 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Renal Cancer; Birt-Hogg-Dube Syndrome
Keywords: Overall Response Rate; Hereditary Cancer Syndrome; mTOR Therapy Naive
MeSH Terms: conditions — Kidney Neoplasms; Birt-Hogg-Dube Syndrome; Neoplastic Syndromes, Hereditary | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Birt-Hogg-Dube Syndrome (Experimental): Birt-Hogg-Dube Syndrome (BHD)-associated renal tumors
  Interventions: Drug: Everolimus
- Sporadic chromophobe renal tumors (Experimental): Sporadic chromophobe renal tumors
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Everolimus is a commercial agent and is supplied by Novartis.

SUMMARY:
Background:

- Research has shown that the drug everolimus can stop cancer cells from growing. It is approved for people with advanced kidney cancer. Researchers want to see if it also helps people with two other types of kidney cancer.

Objective:

- To see if everolimus is safe and effective in people with Birt-Hogg-Dube Syndrome (BHD)-associated kidney cancer or sporadic (nonfamilial) chromophobe renal cancer.

Eligibility:

- People ages 18 and over with BHD-associated kidney cancer or advanced sporadic chromophobe renal cancer.

Design:

* Participants will be screened with:
* Medical history, physical exam, and blood and urine tests.
* Computed tomography (CT) scan or magnetic resonance imaging (MRI) scan. They will lie in a machine that takes pictures of their chest/abdomen/pelvis.
* They may also be screened with:
* Another scan, of the brain or neck.
* Bone scan.
* Positron emission tomography scan with fludeoxyglucose (FDG-PET).
* Heart and lung tests.
* Tests for hepatitis.
* Participants will take a tablet once a day by mouth for up to a year. They will keep a diary of when they take the tablet and any symptoms.
* During the study, participants will have physical exams and urine and blood tests. They will have scans of the chest/abdomen/pelvis. They may have FDG-PET and bone scans.
* Participants will have tests for hepatitis and may have a tumor sample taken.
* Participants will have a follow-up visit 4-5 weeks finishing taking the drug. They will have a physical exam and blood tests. They may have scans and/or hepatitis tests.
* Participants will be called about every 3-6 months after the study ends to see how they are doing

DETAILED DESCRIPTION:
Background:

* Birt-Hogg-Dube (BHD) is a hereditary cancer syndrome with clinical manifestations including cutaneous fibrofolliculomas, lung cysts/pneumothorax, and renal cell carcinoma (RCC). RCC occurs in approximately 30% of patients with BHD. It presents at an early age of onset and is commonly bilateral and multifocal.
* Tumors associated with BHD can have variable histology, however approximately 85% of these tumors have a chromophobe component (either alone or part of a hybrid tumor mixed with elements of oncocytoma).
* The current management includes surgical resection with partial nephrectomy when tumors reach 3 cm. While significant morbidity can be associated with repeat, partial nephrectomy with this approach, most patients can maintain renal function and do not develop systemic disease. There are no proven systemic therapy options for BHD to date.
* Germline mutations in the gene Folliculin (FLCN) are the genetic hallmark of BHD and can be found in greater than 90% of patients. FLCN is believed to function like a classic tumor suppressor gene with a second hit in the wild type allele (somatic mutation or loss of heterozygosity) occurring in the majority of renal tumors.
* BHD is in the family of hamartomatous disorders similar to Tuberous Sclerosis Complex (TSC) and Cowden Syndrome, and studies have found activation of the phosphoinositide 3-kinase (PI3K)/mTOR pathway in BHD renal tumors. FLCN is believed be part of a complex that interacts with 5' AMP-activated protein kinase (AMPK) and is involved with regulation of mTOR activity. In vitro and in vivo models of FLCN loss demonstrate activation of both mTOR complex 1 (mTORC1) and mTOR complex 2 (mTORC2).
* Preclinical data from conditional FLCN knockout mice demonstrate that treatment with sirolimus can reverse renal manifestations.
* We hypothesize that mTOR inhibition with everolimus treatment will be clinically active in BHD associated RCC.

Objectives:

-To determine the overall response rate with everolimus treatment in subjects with BHD-associated renal tumors.

Eligibility:

-Patients with renal cell carcinoma (RCC) associated with Birt-Hogg-Dube Syndrome (BHD).

Design:

* This is an open label, phase II study to evaluate the efficacy and safety of everolimus therapy in patients with BHD associated renal tumors. Up to 16 evaluable patients will be enrolled.
* Tumor response rate will be measured by Response Evaluation Criteria in Solid Tumors (RECIST) and efficacy analysis will be done.
* Secondary endpoints will evaluate growth rates (cm/year) while on therapy.
* Additionally, reduction in the size of lung cysts and cutaneous fibrofolliculomas will be evaluated.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have a clinical diagnosis of Birt-Hogg-Dub (Copyright) Syndrome (clinical features consistent with BHD and /or a germline Folliculin (FLCN) mutation) and the presence of localized, locally advanced or advanced, renal tumor(s).
* Patients must have measurable disease, as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Age greater than or equal to 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1 (Karnofsky greater than or equal to 70%).
* Patients must have normal organ and marrow function as defined below:

leukocytes greater than or equal to 3,000/mcL

absolute neutrophil count greater than or equal to 1,500/mcL

platelets greater than or equal to 100,000/mcL

total bilirubin less than or equal to 2mg/dL

Aspartate aminotransferase (AST) Serum glutamic oxaloacetic transaminase(SGOT)/Alanine aminotransferase (ALT) Serum glutamic pyruvic transaminase(SGPT) greater than or equal to 2.5 times institutional upper limit of normal (ULN) (greater than or equal to 5 times ULN in patients with liver metastases)

creatinine less than or equal to 2.0 times ULN

OR

creatinine clearance greater than or equal to 30 mL/min/1.73 m(2)

fasting serum cholesterol less than or equal to 300 mg/dL OR less than or equal to 7.75 mmol/L

AND

fasting triglycerides less than or equal to 2.5 times ULN

NOTE: In case one or both of these thresholds (for fasting serum cholesterol or triglyceride) are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.

* No history of major bleeding, recent or active myocardial ischemia, gastrointestinal (GI) perforation, cerebrovascular accidents or other significant illness.
* Recovery from acute toxicity of prior treatment for renal cell carcinoma (RCC) (to less than or equal to grade 1 the active version of Common Terminology Criteria for Adverse Events (CTCAE) or to a level permitted under other sections of Inclusion/ Exclusion criteria). Additionally, in patients who have received standard or experimental treatments for their RCC at least approximately 5 half-lives should have elapsed from the last dose at the time of study entry.
* No prior therapy with an mTOR-pathway inhibitor.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients currently receiving anticancer therapies (including chemotherapy, radiation therapy, antibody based therapy, etc.).
* Known intolerance or hypersensitivity to everolimus or other rapamycin analogs (e.g. sirolimus, temsirolimus).
* Patients with known brain metastases unless treated with an appropriate modality with no evidence of progression/recurrence for >3months
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring intravenous (IV) antibiotics, invasive fungal infection, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with everolimus. Known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral everolimus.
* Uncontrolled diabetes mellitus as defined by hemoglobin A1c (HbA1c) >8% despite adequate therapy. Patients with a known history of impaired fasting glucose or diabetes mellitus (DM) may be included, however blood glucose and antidiabetic treatment must be monitored closely throughout the trial and adjusted as necessary.
* Patients who have any severe and/or uncontrolled medical conditions such as:

  1. unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction less than or equal to 6 months prior to start of everolimus, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease.
  2. Symptomatic congestive heart failure of New York heart Association Class III or IV.
  3. known severely impaired lung function (spirometry and diffusing capacity of the lung for carbon monoxide (DLCO) 50% or less of normal and oxygen (O2) saturation 88% or less at rest on room air).
  4. active, bleeding diathesis.
* Chronic (treatment > 1 month) or ongoing treatment with corticosteroids or other immunosuppressive agents. Topical or inhaled corticosteroids are allowed.
* Patients who have received live attenuated vaccines within 1 week of start of everolimus Examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, Bacillus Calmette-Guerin (BCG), yellow fever, varicella and typhoid vaccine) TY21a typhoid vaccines.
* Patients, who in the opinion of the investigator, are unlikely to comply with follow-up visits or other study requirements. Patients who are currently part of or have participated in any clinical investigation with an investigational drug within 1 month prior to dosing.
* Pregnant or nursing (lactating) women.
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, who do not agree to use highly effective methods of contraception during the study and 8 weeks after.

  * Highly effective contraception methods include combination of any two of the following:

    1. Use of oral, injected or implanted hormonal methods of contraception or;
    2. Placement of an intrauterine device (IUD) or intrauterine system (IUS);
    3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository;
    4. Total abstinence or;
    5. Male/female sterilization.

Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to randomization. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential.

* Male patients whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment.
* Prior invasive malignancy of other histology currently requiring treatment.
* Patients with active Hepatitis B (detectable hepatitis B virus-deoxyribonucleic acid (HBV-DNA) or hepatitis B virus surface antigen (HBsAg +) or Hepatitis C infection (detectable hepatitis C virus ribonucleic acid (HCV RNA) by polymerase chain reaction (PCR)
* Patients who are currently on or have used potent or moderate inhibitors or strong inducers Cytochrome P450 3A4 (CYP3A4) or P-glycoprotein (PgP) inhibitors in the past 2 weeks

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2018-04-17 (Actual); Study Completion 2018-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramaprasad Srinivasan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Schmidt LS. Birt-Hogg-Dube syndrome: from gene discovery to molecularly targeted therapies. Fam Cancer. 2013 Sep;12(3):357-64. doi: 10.1007/s10689-012-9574-y. PMID 23108783
- [Background] Birt AR, Hogg GR, Dube WJ. Hereditary multiple fibrofolliculomas with trichodiscomas and acrochordons. Arch Dermatol. 1977 Dec;113(12):1674-7. PMID 596896
- [Background] Schmidt LS, Warren MB, Nickerson ML, Weirich G, Matrosova V, Toro JR, Turner ML, Duray P, Merino M, Hewitt S, Pavlovich CP, Glenn G, Greenberg CR, Linehan WM, Zbar B. Birt-Hogg-Dube syndrome, a genodermatosis associated with spontaneous pneumothorax and kidney neoplasia, maps to chromosome 17p11.2. Am J Hum Genet. 2001 Oct;69(4):876-82. doi: 10.1086/323744. Epub 2001 Aug 30. PMID 11533913

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Sporadic chromophobe renal tumors arm/group is not included here and throughout because the protocol was amended to remove the Sporadic chromophobe renal tumors arm/group. The study was unable to enroll participants with this disease.
Period: Overall Study
Arm/Group | Birt-Hogg-Dube Syndrome
Started | 3
Completed | 1
Not Completed | 2
Not completed — Adverse event-pneumonitis | 2

BASELINE CHARACTERISTICS:
Arm/Group | Birt-Hogg-Dube Syndrome
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (10.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2
  Asian | 1
  A person not meeting definition of Hispanic/Latino | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate With Everolimus Treatment.
Description: Overall best response is defined as the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Response was assessed by the Response Evaluation in Solid Tumors (RECIST) criteria v1.1. Progressive disease is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of at least 5mm. Note: the appearance of one or more new lesions is also progression. Complete response is disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the diameters of target lesions. Stable disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study.
Time Frame: End of treatment: every 12 weeks up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Birt-Hogg-Dube Syndrome
Number analyzed (Participants) | 3
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 3
  Progressive Disease | 0

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival is defined as the time interval from start of treatment to documented evidence of disease progression. Progression is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of at least 5mm. Note: the appearance of one or more new lesions is also progression. Progressive disease was assessed by the Response Evaluation in Solid Tumors (RECIST) criteria v1.1.
Time Frame: median follow-up time: 9 months
Population: Because all the 3 patients were alive without progression as of date of off study their median time to progression cannot be determined.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Birt-Hogg-Dube Syndrome
Number analyzed (Participants) | 3
Months | NA [NA to NA] — Insufficient number of patients with events.

3. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival is defined as the time between the first day of treatment to the day of death.
Time Frame: From the first day of treatment to the day of death, up to 1 year
Population: Because all the 3 patients were alive as of date of off study, their median time to death is unknown.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Birt-Hogg-Dube Syndrome
Number analyzed (Participants) | 3
Months | NA [NA to NA] — Insufficient number of patients with events.

4. Secondary Outcome: Count of Participants With Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence.
Time Frame: Date treatment consent signed to date off study, approximately 8 months and 28 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Birt-Hogg-Dube Syndrome
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 8 months and 28 days.
Arm/Group | Birt-Hogg-Dube Syndrome
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Birt-Hogg-Dube Syndrome (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Cholesterol high (Investigations) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 2 (5)
Dizziness (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Fatigue (Gastrointestinal disorders) | 1 (2)
Headache (Nervous system disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (3)
Hemoglobinuria (Renal and urinary disorders) | 1 (1)
Hyperglycemia (Investigations) | 1 (1)
Hypertriglyceridemia (Investigations) | 3 (6)
Infections and infestations - Other, Upper Respiratory Infection (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Neutrophil count decreased (Investigations) | 1 (9)
Pain (Gastrointestinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 1 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-03-07): https://cdn.clinicaltrials.gov/large-docs/92/NCT02504892/Prot_SAP_000.pdf
  • Informed Consent Form (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/92/NCT02504892/ICF_001.pdf